CLINICAL TRIAL: NCT06625970
Title: A Randomized Phase III Trial With a Factorial Design Evaluating the Efficacy and Safety of Darolutamide and Stereotactic Dose Escalated Radiotherapy in Patients With Localized Prostate Cancer and High-risk Features of Relapse, From the Prostate Cancer Consortium in Europe (PEACE)
Brief Title: Study Evaluating the Efficacy and Safety of Darolutamide and Stereotactic Dose Escalated Radiotherapy in Patients With Localized Prostate Cancer and High-risk Features of Relapse
Acronym: PEACE 7
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UC-GTG-2310; 2023-509787-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: High Risk Prostate Carcinoma; Prostate Cancer
Keywords: HPRC, PSMA-PET, Prostate Cancer, High-Risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Radiosurgery; Androgen Antagonists; Standard of Care; Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1:1:1) to receive either:
  * Arm A (Standard arm): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy
  * Arm B (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy + darolutamide
  * Arm C (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT
  * Arm D (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT + darolutamide
  Patients will be stratified according to the number of risk factors (2 vs. 3) and the presence of a dominant intraprostatic lesion prostate imaging-reporting and data system (PI-RADS) 5 (yes vs no) and investigational site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Standard arm) (Other): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy
  Interventions: Drug: ADT (Standard of Care); Radiation: radiotherapy
- Arm B (Experimental arm): (Experimental): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy + darolutamide
  Interventions: Drug: Darolutamide; Drug: ADT (Standard of Care); Radiation: radiotherapy
- Arm C (Experimental arm): (Experimental): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT
  Interventions: Radiation: Stereotactic Body RadioTherapy (SBRT); Drug: ADT (Standard of Care); Radiation: radiotherapy
- Arm D (Experimental arm): (Experimental): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT + darolutamide
  Interventions: Drug: Darolutamide; Radiation: Stereotactic Body RadioTherapy (SBRT); Drug: ADT (Standard of Care); Radiation: radiotherapy

INTERVENTIONS:
Drug: Darolutamide — Pharmaceutical form: 300 mg tablets Administration route: oral (PO) Posology: 600 mg twice daily (BID)
  Arms: Arm B (Experimental arm):; Arm D (Experimental arm):
Radiation: Stereotactic Body RadioTherapy (SBRT) — Following randomization, patients will receive dose escalated intensity modulated radiotherapy (IMRT) using normo-fractionation or moderate hypo-fractionation including whole pelvic nodal radiotherapy (WPRT).
  At study entry, each investigational site will be asked to choose one regimen (normo-fractionation or moderate hypo-fractionation) which will be applied for all patients included by the investigational site in the study.
  SBRT, experimental treatment, will be used as a boost in Arms C & D. The placement of 3 to 4 fiducial markers for stereotactic boost is mandatory.
  SBRT will be applied only on Prostate: 2 times 10 Gy delivered to the prostate with a gap of one week between each SBRT fraction.
  Arms: Arm C (Experimental arm):; Arm D (Experimental arm):
Drug: ADT (Standard of Care) — Androgen Deprivation Therapy (ADT)
  The ADT treatment will be chosen at the investigator's discretion, and will be administered according to local standard procedures for up to 2 years.
  Patients who may have received ADT prior joining the study should have started the ADT treatment within a maximum of 6 weeks before randomization. Otherwise ADT will be started on Day 1 (or 14 days at the latest after the randomization).
  Other Names: LHRH agonists; LHRH antagonists
Radiation: radiotherapy — Following randomization, patients will receive dose escalated intensity modulated radiotherapy (IMRT) using normo-fractionation or moderate hypo-fractionation including whole pelvic nodal radiotherapy (WPRT).
  Arm A and Arm B:
  If Normo-fractionated radiotherapy: Pelvic nodes 46 Gy, seminal vesicles 46-54 Gy and prostate 78 Gy (39 fractions over 8 weeks).
  If Hypo-fractionated radiotherapy: Pelvic nodes and seminal vesicles 44 Gy in 20 fractions; prostate 60 Gy delivered concomitantly in 20 fractions over 4 weeks.
  Arm C and Arm D:
  If Normo-fractionated radiotherapy: Pelvic nodes 46 Gy, seminal vesicles 46 Gy in 23 fractions over 4.5 weeks.
  If Hypo-fractionated radiotherapy: Pelvic nodes and seminal vesicles 44 Gy in 20 fractions over 4 weeks.
  Other Names: Normo-fractionated radiotherapy; Hypo-fractionated radiotherapy; intensity modulated radiotherapy (IMRT); whole pelvic nodal radiotherapy (WPRT)

SUMMARY:
PEACE 7 is an international, multicenter, randomized, open-label phase III study that aims at evaluating the efficacy and safety of darolutamide and of stereotactic dose escalated prostate radiotherapy in patients with localised prostate cancer and high-risk features of relapse (defined as patients with at least 2 high-risk criteria from National Comprehensive Cancer Network (NCCN) classification) using a factorial (2x2) design.

The primary objective of this study is to assess the efficacy of darolutamide and of a stereotactic dose escalated radiotherapy targeting prostate in combination with ADT and pelvic nodal radiotherapy in terms of metastasis-free survival (MSF).

Patients will be randomized (1:1:1:1) to receive either:

* Arm A (Standard arm): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy
* Arm B (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated prostate radiotherapy including pelvic nodal radiotherapy + darolutamide
* Arm C (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT
* Arm D (Experimental arm): ADT + conventional fractionated or moderately hypo-fractionated pelvic nodal radiotherapy + Prostate SBRT + darolutamide

Patient will receive systemic treatments (ADT and/or darolutamide) during 2 years where visits on site are planned at D45, D90, D180 and then every 3 months for checkups and follow prostate specific antigen (PSA) level.

Metastasis-free survival (MFS) is defined as the time interval from randomization to the date of the appearance of metastasis (on next generation imaging) or death (from any cause), whichever occurs first. Radiographic evaluation will be carried out at the time of biochemical failure (Phoenix criteria) or in case of clinical suspicion. After biochemical failure (Phoenix criteria) radiographic evaluation on next generation imaging (prostate-specific membrane antigen (PSMA) positron emission tomography (PET) scan (any European Medicines Agency (EMA) approved PSMA tracer)) will be performed every 6 months until a metastatic site of relapse is identified and will be repeated at each subsequent PSA progression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures

   Note: In case of physical incapacitation, a trusted representative of their choice, which is not the investigator or sponsor, can sign on the behalf of the patients
2. Men, 18 years ≤ Age ≤ 80 years
3. ECOG performance status of 0 or 1
4. No significant co-morbidities that might prevent long-term follow-up
5. Histologically confirmed adenocarcinoma of the prostate
6. Meet at least 2 of the following criteria from NCCN classification:

   * Gleason score ≥8
   * T3 or T4 disease (T3 defined by MRI is acceptable)
   * Prostate-specific antigen ≥20 ng/mL
7. Prostate size on MRI <100 cc
8. Absolute neutrophil count ≥ 1.5 x 10⁹/L
9. Platelet count ≥100 x 10⁹/L
10. Haemoglobin ≥90 g/L (in absence of red blood cell transfusion within 4 weeks prior to randomization)
11. Hepatic function: serum alanine aminotransferase (ALT) and/or aspartate transaminase (AST) ≤2.5 x upper limit of normal (ULN), total bilirubin ≤1.5 x ULN
12. Creatinine ≤2.0 x ULN
13. Sexually active patients must agree to use an effective contraceptive method while on treatment and for 1 week after the final dose of investigational product
14. Patient must be affiliated to a Social Security System or in possession of equivalent private health insurance (according to local regulations for participation in clinical trials)
15. Patient must be willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits, and examinations including follow-up

Exclusion Criteria:

1. Clinically or radiologically detectable metastasis, including no evidence of pelvic lymph node metastasis on next generation imaging (PSMA PET/CT), nor enlarged pelvic lymph nodes (≥1 cm in small diameter) on MRI Note: Patients with infra-centimetric nodal disease (<1 cm in small diameter) on conventional imaging and equivocal hyperfixation on next generation imaging may be included
2. Recent history of TURP or prostate enucleation (less than 6 months) Note: patients with severe obstructive symptoms (defined as International Prostate Symptom Score (IPSS) ≥20) should be carefully evaluated to rule out the need for TURP/Prostate enucleation
3. Prior treatment for prostate cancer, including prostatectomy, except lymph node dissection (patients with PN- disease only can be accrued) or ADT (started more than 6 weeks before randomization)
4. Patient with other known concurrent severe and/or uncontrolled concurrent medical disease or infection (such as active viral hepatitis, active human immunodeficiency virus (HIV) or chronic liver disease) or co-morbidity, which could compromise participation in the study
5. Cardiac disease such as uncontrolled hypertension (systolic BP ≥160 mmHg or diastolic BP ≥95 mmHg; 3 consecutive measures taken 5 minutes apart), stroke, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within one year, coronary/peripheral artery bypass graft, LVEF > grade 2
6. Uncontrolled diabetes mellitus
7. Current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, stable chronic liver disease per investigator assessment)
8. Gastrointestinal disorder or procedure, which expects to interfere significantly with absorption of study treatment. Severe GI disorders precluding pelvic irradiation
9. Known severely impaired lung function (spirometry and DLCO 70% or less of normal and O2 saturation of 88% or less at rest on room air)
10. Other prior malignancy within the last 3 years, except basal cell skin cancer
11. Known hypersensitivity to the study treatment or any of its ingredients.
12. Physical or psychological condition or any condition that in the opinion of the investigator would impair the patients' ability to comply with the study procedures
13. Previous treatment for prostate cancer (surgery or radiotherapy) or previous pelvic irradiation that would make prostate/pelvis radiotherapy impossible
14. Concomitant prohibited treatment. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5. A one-week washout period is necessary for patients who are already on these treatments
15. Prior treatment with second generation androgen receptor (AR) inhibitors, other investigational AR inhibitors, or CYP17 enzyme inhibitor
16. Use of oestrogens or 5-α reductase inhibitors or AR inhibitors
17. Acute toxicities of prior treatments and procedures not resolved to grade ≤1 or baseline before randomization
18. Prior chemotherapy or immunotherapy for prostate cancer
19. Major surgery within 28 days before randomization
20. Participation in another therapeutic trial within 30 days prior to inclusion
21. Persons deprived of their liberty or under protective custody or guardianship
22. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2045-10 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | from randomization to the onset of metastasis or death, up to 8.5 years
  Metastasis-free survival (MFS) is defined as the time interval from randomization to the date of the appearance of metastasis (on next generation imaging) or death (from any cause), whichever occurs first.

SECONDARY OUTCOMES:
Clinical Progression-Free Survival | From randomization to disease progression, up to 8.5 years
  Clinical Progression-Free Survival (cPFS) is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. Clinical disease progression is defined as metastatic relapse or proven local relapse (by either biopsy or unequivocal imaging), unequivocal nodal progression on imaging, or death (from any cause), whichever occurs first.
Biochemical Progression-Free Survival | From randomization to PSA relapse or death, up to 8.5 years
  Biochemical Progression-Free Survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse. Biological disease progression is defined as the time interval from randomization to the date of PSA relapse or death (from any cause), whichever occurs first.
Time to local relapse | From randomization to local disease progression, up to 8.5 years
  Time to local relapse is defined as the time interval from randomization to the date of the appearance of the first proven local relapse (by either biopsy or unequivocal imaging).
Prostate Cancer-Specific Survival (PCSS) | From randomization to death due to prostate cancer, up to 8.5 years
  Prostate Cancer-Specific Survival (PCSS) is defined as the time interval between randomization and the date of death due to prostate cancer.
Overall Survival (OS) | From randomization to death, up to 20 years
  Overall Survival (OS) is the length of time from randomization that patients enrolled in the study are still alive

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Pierre BLANCHARD, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Gilles CREHANGE, MD, PhD, Study Chair — Institut Curie
Locations (6):
- France (5):
  - Clinique Pasteur Lanroze - Brest, Brest
  - Centre Georges Francois Leclerc, Dijon
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - CHU Saint-Etienne, Saint-Etienne
  - Gustave Roussy, Cancer Campus, Grand Paris, Villejuif
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients